CLINICAL TRIAL: NCT05140200
Title: An Open-label, Single Dose Study to Investigate the Pharmacokinetics, Safety, Tolerability and Immunogenicity of Two Dose Levels of GSK3511294 Administered Subcutaneously in Chinese Healthy Participants
Brief Title: Study of GSK3511294 in Healthy Chinese Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 208021
Record Dates: First submitted 2021-11-22; First posted 2021-12-01 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Asthma
Keywords: Single dose study; Immunogenicity; GSK3511294; Chinese healthy participants
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Masking Description: This is an open-label study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1: Participants receiving GSK3511294 at Dose level 1 (Experimental)
  Interventions: Biological: GSK3511294
- Cohort 2: Participants receiving GSK3511294 at Dose level 2 (Experimental)
  Interventions: Biological: GSK3511294

INTERVENTIONS:
Biological: GSK3511294 — GSK3511294 will be administered.

SUMMARY:
This single dose pharmacokinetic (PK) study aims to investigate the PK, safety, tolerability and immunogenicity of two dose levels of GSK3511294 administered subcutaneously in Chinese healthy participants

ELIGIBILITY:
Inclusion Criteria:

* Participant between 18 to 45 years of age.
* Participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, electrocardiograms and vital signs.
* Body weight greater than or equal to (>=)50.0 kilograms (kg) for males, >=45.0 kg for females, and body mass index (BMI) within the range (19.0-26.0) kg/meter square (m^2) (inclusive).
* Contraceptive use by men and/or women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
* Capable of giving signed informed consent.

Exclusion Criteria:

* Participant is pregnant, breastfeeding, or a woman of childbearing potential
* History or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs
* Participants with allergy/intolerance to a monoclonal antibody or biologic or participants with a previous history of clinically significant multiple or severe allergic reactions/intolerance
* Current evidence or recent history of an infective illness
* A positive pre-study drug/alcohol screen or a history (or suspected history) of alcohol misuse or substance abuse
* Clinically significant abnormalities
* Participants with Coronavirus Disease-2019 (COVID-19)
* With prior/concurrent clinical study experience.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2021-12-10 (Actual); Primary Completion 2022-12-23 (Actual); Study Completion 2022-12-23 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curve (AUC) from time zero (pre-dose) extrapolated to infinite time (AUC[0-infinity]) of GSK3511294 | Up to Week 26
AUC from time 0 (pre-dose) to last time of quantifiable concentration within a participant across all treatments (AUC[0-t]) of GSK3511294 | Up to Week 26
AUC from time 0 to Week 4 (AUC[0-Week 4]) of GSK3511294 | Up to Week 4
AUC from time 0 to Week 12 (AUC[0-Week 12]) of GSK3511294 | Up to Week 12
AUC from Time 0 to Week 26 [AUC(0-Week 26)] of GSK3511294 | Up to Week 26
Percentage of AUC(0-infinity) obtained by extrapolation (%AUCex) of GSK3511294 | Up to Week 26
Maximum observed plasma concentration (Cmax) of GSK3511294 | Up to Week 26
Time of occurrence of Cmax (tmax) of GSK3511294 | Up to Week 26
Time to last quantifiable concentration (tlast) of GSK3511294 | Up to Week 26
Apparent clearance (CL/F) of GSK3511294 | Up to Week 26
Apparent volume of distribution (Vz/F) of GSK3511294 | Up to Week 26
Terminal elimination rate constant (lambda z) of GSK3511294 | Up to Week 26
Terminal phase half-life (t1/2) of GSK3511294 | Up to Week 26

SECONDARY OUTCOMES:
Number of participants with adverse events (AEs) and serious adverse events (SAEs) | Up to Week 30
Change from Baseline in platelet count, white blood cell (WBC) count, basophils, eosinophils, lymphocytes, monocytes and neutrophils (10^9 cells per liter) | Baseline (Pre-dose on Day 1) and up to Week 26
Change from Baseline in Red blood cell (RBC) count (10^12 cells per liter) | Baseline (Pre-dose on Day 1) and up to Week 26
Change from Baseline in Hemoglobin (Grams per liter) | Baseline (Pre-dose on Day 1) and up to Week 26
Change from Baseline in hematocrit (Proportion of RBC in blood) | Baseline (Pre-dose on Day 1) and up to Week 26
Change from Baseline in mean corpuscular volume (Femtoliters) | Baseline (Pre-dose on Day 1) and up to Week 26
Change from Baseline in mean Corpuscular Hemoglobin (Picograms) | Baseline (Pre-dose on Day 1) and up to Week 26
Change from Baseline in percentage of Reticulocytes (Percentage of reticulocytes) | Baseline (Pre-dose on Day 1) and up to Week 26
Change from Baseline in Sodium, potassium, calcium, Blood urea nitrogen (Millimoles per liter) | Baseline (Pre-dose on Day 1) and up to Week 26
Change from Baseline in Creatinine, total bilirubin, direct bilirubin (Micromoles per liter) | Baseline (Pre-dose on Day 1) and up to Week 26
Change from Baseline in Alkaline Phosphate (ALP), Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST), Gamma Glutamyl Transferase (GGT) (International units per liter) | Baseline (Pre-dose on Day 1) and up to Week 26
Change from Baseline in Albumin, Total Protein (Grams per liter) | Baseline (Pre-dose on Day 1) and up to Week 26
Absolute values of Complement (C) 3 and C4 | Up to Week 26
Ratio to Baseline of C3 and C4 | Baseline (Pre-dose on Day 1) and up to Week 26
Change from Baseline in systolic and diastolic blood pressure (Millimeters of Mercury) | Baseline (Pre-dose on Day 1) and up to Week 26
Change from Baseline in body temperature (Degrees Celsius) | Baseline (Pre-dose on Day 1) and up to Week 26
Change from Baseline in pulse rate (Beats per minute) | Baseline (Pre-dose on Day 1) and up to Week 26
Change from Baseline in PR Interval, QRS Duration, QT Interval, Corrected QT Interval Using Fridericia's Formula (QTcF) (Milliseconds [msec]) | Baseline (Pre-dose on Day 1) and up to Week 26
Number of participants with positive Anti-drug Antibodies (ADAs) against GSK3511294 | Up to Week 26
Titers of ADA against GSK3511294 | Up to Week 26

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Hangzhou, China

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, a key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com